CLINICAL TRIAL: NCT03472599
Title: Long Term Genital Nerve Stimulation to Improve Urinary Continence
Brief Title: Chronic Electrical Stimulation to Reduce Bladder Hyperreflexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Syracuse VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2512-R; RX002512 (Other Grant/Funding Number: VA Office of Research and Development)
Record Dates: First submitted 2018-03-05; First posted 2018-03-21 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Neurogenic Bladder Dysfunction
Keywords: Neurogenic bladder dysfunction; Genital Nerve Stimulation; Electrical Stimulation; Urinary Incontinence; Spinal cord injury
MeSH Terms: conditions — Urinary Incontinence; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: All subjects will take home skin surface electrodes and a simple one-channel electrical stimulators appropriate for extended use set to the stimulus parameters found effective during an initial urodynamics test. Genital nerve stimulation will be applied either continuously or on-demand when individuals turn stimulation on when they feel the onset of bladder leaking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Genital Nerve Stimulation (Experimental): Study participants in this arm will use take-home genital nerve stimulation for 24+ months in order to assess its effectiveness at decreasing urinary incontinence. In order to set effective genital nerve stimulation parameters, study participants will undergo clinical urodynamics every 6 months in which sensitivity to and tolerance of electrical stimulation are assessed.
  Interventions: Other: Genital Nerve Stimulation

INTERVENTIONS:
Other: Genital Nerve Stimulation — Genital nerve stimulation activates sensory afferents that travel through the pudendal nerves and enters the spinal cord through the sacral dorsal root ganglia. Inhibitory spinal reflex pathways are activated, causing increased sympathetic outflow through the inferior mesenteric ganglion and hypogastric nerve and also decreased parasympathetic efferent drive through the pelvic nerve, resulting in inhibited bladder contractions.

SUMMARY:
Bladder spasms after spinal cord injury (SCI) can result in incontinence, urinary tract infections, kidney damage, trigger dangerous increases in blood pressure and decrease independence and quality of life. The investigators' long-term goal is to develop and provide a "bladder pacemaker" able to restore bladder continence for Veterans with SCI. Electrical stimulation of sensory nerves can stop bladder spasms during a doctor visit. However, this approach has not been tested during long term home use. This proposal will 1) determine how well sensory stimulation reduces incontinence and improves quality of life for Veterans with SCI during 1 year of home use, and 2) produce an effective take home system that can be used by more Veterans and other VAs.

DETAILED DESCRIPTION:
The clinical problem of neurogenic detrusor overactivity (bladder hyper-reflexia) is among the most serious problems encountered by Veterans with neurologic injuries such as spinal cord injury (SCI). The majority of persons with SCI suffer from neurogenic bladder (73%) and only 17% of persons with traumatic SCI manage their bladders with voluntary micturition. The investigators' long-term goal is to develop and clinically implement a "bladder pacemaker" able to restore bladder continence for Veterans with spinal cord injury (SCI). This proposal will 1) determine the long-term effectiveness of genital nerve stimulation (GNS) to chronically ( 1 year) reduce urinary incontinence and improve quality of life for Veterans with SCI, and 2) develop and produce an effective take home GNS system that can be used by more Veterans, given to Veterans at the end of the study and used in future multi-VA studies.

The rationale for studying chronic GNS is based on the demonstration in humans with SCI that abnormal hyper-reflexive bladder contractions can be acutely inhibited and bladder capacity acutely increased using GNS. The peripheral and easily accessible location of the dorsal genital nerve (DGN) allows surface stimulation and therefore provides the potential for a less complicated surgical intervention than is currently available, increasing the number of individuals who could benefit from bladder control neural prostheses. While GNS has been demonstrated to be effective acutely by multiple groups, relatively few groups have attempted to test this approach for more than a day.

ELIGIBILITY:
Inclusion Criteria:

* Suprasacral neurogenic bladder following spinal cord injury, stroke, or multiple sclerosis
* Neurologically stable
* Skeletally mature, over 18 years of age.
* Reflex bladder contractions confirmed by cystometrogram
* At least six (6) months post spinal cord injury, stroke, or multiple sclerosis diagnosis
* Able to understand and comply with study requirements
* Able to understand and give informed consent

Exclusion Criteria:

* Active sepsis
* Open pressure sores on penis
* Significant trauma, erosion or stricture of the urethra
* Pregnancy
* Individuals who do not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Incontinence | Collected over 24 months
  The investigators will collect a record of leakage episodes (metric for incontinence) from the specified period.

SECONDARY OUTCOMES:
Bladder Capacity | Collected over 24 months
  The investigators will measure bladder capacity in mL during acute urodynamics trials

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Gustafson, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (2):
- United States (2):
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourbeau DJ, Creasey GH, Sidik S, Brose SW, Gustafson KJ. Genital nerve stimulation increases bladder capacity after SCI: A meta-analysis. J Spinal Cord Med. 2018 Jul;41(4):426-434. doi: 10.1080/10790268.2017.1281372. Epub 2017 Feb 15. PMID 28198657
- [Result] Bourbeau DJ, Gustafson KJ, Brose SW. At-home genital nerve stimulation for individuals with SCI and neurogenic detrusor overactivity: A pilot feasibility study. J Spinal Cord Med. 2019 May;42(3):360-370. doi: 10.1080/10790268.2017.1422881. Epub 2018 Jan 15. PMID 29334338